CLINICAL TRIAL: NCT01475994
Title: Pilot Study to Assess the Effect of Pollen Challenges in an Environmental Challenge Chamber on Dermal Symptoms in Patients With Atopic Dermatitis
Brief Title: Effect of Pollen Challenges on Dermal Symptoms in Patients With Atopic Dermatitis
Acronym: Neurop
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Collaborators: Hannover Medical School (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 11-01 Neurop
Record Dates: First submitted 2011-11-04; First posted 2011-11-22 (Estimated); Last update posted 2012-04-05 (Estimated); Status verified 2012-04

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Challenge with grass pollen (Experimental)
  Interventions: Other: Grass pollen : Dactylis glomerata
- Challenge with clean air (Placebo Comparator)
  Interventions: Other: Challenge with clean air

INTERVENTIONS:
Other: Grass pollen : Dactylis glomerata — The subjects will be challenged for 4 hours on two consecutive days (Day 1 and Day 2) with either 4000 pollen grains/m3 of dactylis glomerata pollen.
  Arms: Challenge with grass pollen
Other: Challenge with clean air — The subjects will be challenged for 4 hours on two consecutive days (Day 1 and Day 2) with clean air.
  Arms: Challenge with clean air

SUMMARY:
This is a mono-center, randomized, double-blind, placebo-controlled, parallel-group study to assess the effect of challenges with dactylis glomerata pollen in an environmental challenge chamber on dermal symptoms in patients suffering from atopic dermatitis.

After each challenge session and on Day 3, Day 4, and Day 5 blood samples will be taken for biomarker assessments. The severity of atopic dermatitis will be rated with the "SCORing Atopic Dermatitis" (SCORAD), with the objective SCORAD and with the assessment of itch and sleeplessness referring to the past 24 hours by a blinded observer (trained dermatologist) on each day including baseline assessments.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, aged 18-65 years. Women will be considered for inclusion if they are: Not pregnant, as confirmed by pregnancy test (see flow chart) and not nursing. Of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit). Of childbearing potential and using a highly effective method of contraception during the entire study (vasectomised partner, sexual abstinence - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the first dose of study medication until at least 72 hours after the last pollen challenge -, implants, injectables, combined oral contraceptives, hormonal IUDs or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap).
* Positive IgE level for Dactylis glomerata of at least CAP FEIA class 3.
* atopic dermatitis (AD) fulfilling the UK criteria of AD
* SCORAD between 20 and 50 points.
* forced Expiratory Volume in the first second (FEV1) ≥ 80% pred. at screening.
* Smokers or non-smokers.
* Body Mass Index ≥18 and ≤ 35.

Exclusion Criteria:

* • Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease.
* Asthma other than mild asthma which is treated with short acting beta-2-agonists only and which is controlled according to the current GINA guidelines
* Clinically relevant abnormalities in haematology, blood chemistry, or urinalysis at screening.
* Positive HIV-1/2Ab, hepatitis B surface antigen (HBsAg) or hepatitis C virus antibodies (HCV-Ab) test at screening.
* Treatment with medication that might interfere with rescue medication for anaphylactic reactions (e.g. beta blocker).
* Topical steroid treatment (wash out phase: 2 weeks)
* Topical calcineurin inhibitor treatment (wash out phase 2 weeks)
* UV radiation treatment (wash out phase 4 weeks)
* Systemic immunosuppression treatment (steroids, cyclosporine, azathioprine, Mycophenolat Mofetil (MMF); wash out phase 4 weeks)
* Treatment with antihistamines (wash out phase 1 week)
* Unstable AD during Screening (SCORAD difference of >10 points from Visit 1 to Visit 2)
* Diastolic blood pressure above 95 mmHg.
* Febrile illness within 2 weeks prior to screening.
* Alcohol or drug abuse within 12 month prior to screening.
* Regular daily consumption of more than 1 liter of usual beer or the equivalent quantity of approximately 40 g of alcohol in another form.
* Participation in another clinical trial 30 days prior to enrolment.
* There is a risk of non-compliance with study procedures.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
SCORAD | Day 1/Baseline vs. Day 3
  Change in SCORAD between Day 1/ baseline (assessed 60 minutes prior to challenge) and Day 3 (assessed post-challenge)

SECONDARY OUTCOMES:
SCORAD Day 4 and 5 | Day 1/Baseline vs. Day 4 and 5
  Change in SCORAD between Day 1 (assessed 60 minutes prior to challenge) and the Scorad on Day 4 and Day 5 (assessed post challenge).

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, MD, professor, Principal Investigator — The Fraunhofer-Gesellschaft